CLINICAL TRIAL: NCT04728022
Title: Brain Research Apprenticeships in New York at Columbia (BRAINYAC)
Brief Title: Brain Research Apprenticeships in New York at Columbia
Acronym: BRAINYAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAT4760; 1R25NS115551-01 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Educational Activities
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: All students in the study will be in the same group, as it is a pre-post measurement based on a summer mentored high school program. Findings will be supplemented with focus groups and interviews.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students (Experimental): Education program
  Interventions: Behavioral: Education program

INTERVENTIONS:
Behavioral: Education program — Mentored high school summer research program

SUMMARY:
The objective of the BRAINYAC program is to prepare high school students for, and deliver, the experience of working in a neuroscience research laboratory over a summer. Our program goals are to prepare local students from Upper Manhattan and the South Bronx with the skills necessary to enter a working research laboratory over a period of 8 months, and support them in learning key laboratory skills and communicating them to an audience.Our hypothesis is that students' self-reports of scientific effectiveness and science identity will improve over the course of the 8-month long program. Self-reported efficacy measures predict academic performance in science, so an improvement in these self-report measures may indicate a higher likelihood to succeed in science, technology, engineering and math (STEM) studies or careers. Likewise, science identity has a positive impact on a student's likelihood of entering a science career, particularly in populations that are under-represented in science.Over a 4-year period we will track students' self-reports of (1) scientific efficacy, including their level of confidence in scientific writing, oral presentation, library and literature search, conducting research and general academic skills, and (2) science identity. We will adopt a mixed-methods approach combining survey data with focus groups and interviews to present a full picture of these changes. We also propose to track students after they leave the program, to measure whether the changes in scientific self-efficacy translate into STEM studies at the level of higher education or career choices. We will also obtain data from scientific mentors in the program to inform us whether we are adequately supporting them in providing the students with training.

DETAILED DESCRIPTION:
This study will utilize a mixed methodological approach integrating quantitative and qualitative data elements. It will employ a one-group, pretest-posttest research design, in order to allow us to determine the effect of participation in the BRAINYAC program (i.e., the intervention) on participating students' STEM development (i.e., efficacy and identity). The study will also include retrospective individual and focus group interviews in order to obtain a fuller understanding of the concepts under study (e.g., scientific identity, readiness to pursue science, etc.) from the students' point of reference. To the extent possible, the study will incorporate a longitudinal analysis in order to examine how program participation affects students' academic and career decisions in their final high school and postsecondary years through retrospective surveys of alumni participants. In addition to assessing program impact, the research design will include an evaluation component to examine program implementation. Through an examination of program documentation (e.g., student attendance, descriptions of activities) and retrospective surveys of participants (i.e., students and mentors) this component will determine the extent to which the program was implemented as proposed. It will provide valuable information connecting program elements to observed outcomes and can be used to make modifications to the research and/or program designs, as needed.

ELIGIBILITY:
Inclusion Criteria:

* All students and mentors in the program will be invited to enroll

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Self-report of scientific effectiveness | 8 months
  Change in Likert score
Self-report of scientific identity | 8 months
  Change in Likert score
Likelihood of studying science in college or going on to a science career | 4 years
  Change in Likert score

CONTACTS AND LOCATIONS:
Overall Officials: Daphna Shohamy, PhD, Principal Investigator — Columbia University
Locations (1):
- Zuckerman Institute, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Program web page — https://zuckermaninstitute.columbia.edu/brainyac